CLINICAL TRIAL: NCT03438344
Title: A Phase II Randomized, Placebo-Controlled, Multicenter Trial to Evaluate the Protective Function of a CMV-MVA Triplex Vaccine in Recipients of a Haploidentical Hematopoietic Stem Cell Transplant
Brief Title: Multi-antigen CMV-Modified Vaccinia Ankara Vaccine in Reducing CMV Related Complications in Patients With Blood Cancer Undergoing Donor Stem Cell Transplant
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI Withdrawal
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 17366
Record Dates: First submitted 2017-12-29; First posted 2018-02-19 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Acute Lymphoblastic Leukemia in Remission; Acute Myeloid Leukemia in Remission; Bone Marrow Transplantation Recipient; Chronic Lymphocytic Leukemia; Chronic Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Hematopoietic Cell Transplantation Recipient; Hodgkin Lymphoma; Myelodysplastic Syndrome; Myelofibrosis; Myeloproliferative Neoplasm; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Chronic-Phase; Hodgkin Disease; Myelodysplastic Syndromes; Primary Myelofibrosis; Myeloproliferative Disorders; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (CMV-MVA triplex vaccine) (Experimental): Patients receive multi-antigen CMV-modified vaccinia Ankara vaccine via injection on days 28 and 56 post-HCT.
  Interventions: Biological: Multi-antigen CMV-Modified Vaccinia Ankara Vaccine; Other: Laboratory Biomarker Analysis
- Arm II (placebo) (Placebo Comparator): Patients receive placebo via injection on days 28 and 56 post-HCT.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo

INTERVENTIONS:
Biological: Multi-antigen CMV-Modified Vaccinia Ankara Vaccine — Given IM
  Other Names: CMV-MVA Triplex Vaccine
  Arms: Arm I (CMV-MVA triplex vaccine)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo — Given IM
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)

SUMMARY:
This randomized phase II trial studies how well multi-antigen cytomegalovirus (CMV)-modified vaccinia Ankara vaccine works in reducing CMV related complications in patients with blood cancer who are undergoing donor stem cell transplant. Vaccines made from a gene-modified virus may help the body build an effective immune response to kill cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if multi-antigen CMV-modified vaccinia Ankara vaccine (CMV-modified vaccinia Ankara [MVA] triplex) reduces the frequency of CMV events, defined as reactivation or CMV disease in CMV+, haploidentical hematopoietic cell transplantation (haploHCT) recipients.

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of CMV-MVA triplex in vaccinated, haploHCT recipients by assessing the following: non-relapse mortality (NRM) at 100 days post hematopoietic cell transplantation (HCT), severe (grade 3-4) acute graft versus host disease (GVHD), and grade 3-4 adverse events (AEs) probably or definitely related to the vaccination within 2 weeks from each vaccination.

II. To characterize CMV related events in recipients of CMV-MVA triplex compared to placebo, by assessing time to viremia (number of days from transplantation to the date of >= 1250 IU/mL), duration of viremia, recurrence of viremia, incidence of late CMV viremia/disease (> 100 and =< 360 days post HCT), use of antiviral drugs (triggered by clinically significant viremia of >= 1250 IU/mL), cumulative number of CMV specific antiviral treatment days.

III. To evaluate the impact of CMV-MVA triplex on transplant related outcomes by assessing the incidence of acute graft versus host disease (aGVHD), chronic GVHD, relapse, non-relapse mortality, all-cause mortality, infections.

IV. To determine if CMV-MVA triplex increases levels, function and kinetics of CMV-specific T cell immunity in vaccinated compared to placebo treated, CMV seropositive HCT-recipients.

V. To determine whether vaccination induces adaptive natural killer (NK) cell population changes, and increase in the highly cytotoxic memory NKG2C+ NK cell.

VI. To compare GVHD biomarkers between the vaccine and placebo groups.

OUTLINE: Patients are randomized into 1 of 2 arms.

ARM I: Patients receive multi-antigen CMV-modified vaccinia Ankara vaccine intramuscularly (IM) on days 28 and 56 post-HCT.

ARM II: Patients receive placebo IM on days 28 and 56 post-HCT.

After completion of study treatment, patients are followed up at 100, 140, 180, 270, and 365 days, and then periodically for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have the ability to understand and the willingness to sign a written informed consent
* Participant must be willing to comply with study and/or follow-up procedures, including willingness to be followed for one year post-HCT
* Planned peripheral blood stem cell (PBSC) or bone marrow (BM) HCT for the treatment of the following hematologic malignancies:

  * Lymphoma (Hodgkin and non-Hodgkin)
  * Myelodysplastic syndrome
  * Acute lymphoblastic leukemia in first or second remission (for acute lymphoblastic leukemia/lymphoblastic lymphoma, the disease status must be in hematologic remission by bone marrow and peripheral blood; persistent lymphadenopathy on computed tomography [CT] or CT/positron emission tomography [PET] scan without progression is allowed)
  * Acute myeloid leukemia in first or second remission
  * Chronic myelogenous leukemia in first chronic or accelerated phase, or in second chronic phase
  * Other hematologic malignancies judged appropriate by the clinical principal investigators (PIs), including chronic lymphocytic leukemia, myeloproliferative disorders and myelofibrosis; patients with multiple myeloma and those with non-malignant disease such as aplastic anemia are excluded

    * Adult cases of multiple myeloma (MM) are excluded; adults with aplastic anemia are excluded; patients undergoing a second haploHCT are not eligible (patients who have undergone a previous autologous HCT are eligible)
* Patients receiving myeloablation (MA) or reduced intensity conditioning (RIC) are allowed
* CMV seropositive (recipient)
* Planned related HCT with molecular 3/6 (haploidentical) intermediate/high resolution human leukocyte antigen (HLA) donor allele matching
* Planned HCT with minimal to no-T cell depletion of graft
* Conditioning and immunosuppressive regimens according to institutional guidelines are permitted
* Negative serum or urine beta-human chorionic gonadotropin (HCG) test (female patient of childbearing potential only) within two weeks of registration
* Seronegative for human immunodeficiency virus (HIV), hepatitis C virus (HCV) and active hepatitis B virus (HBV) (surface antigen negative) within 2 months of registration and no history of disseminated cutaneous human papillomavirus (HPV) related disease
* Agreement by females of childbearing potential and sexually active males to use an effective method of contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for up to 90 days post-HCT; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately

Exclusion Criteria:

* Any prior investigational CMV vaccine
* Experimental anti-CMV chemotherapy in the last 6 months
* Live attenuated vaccines
* Medically indicated subunit (Engerix-B for HBV, Gardasil for HPV) or killed vaccine (e.g. influenza, pneumococcal, or allergy treatment with antigen injections)
* Allergy treatment with antigen injections
* Alemtuzumab or any equivalent in vivo T-cell depleting agent (or CD34+ selection)
* Antiviral medications with known therapeutic effects on CMV such as ganciclovir/valganciclovir (GCV/VAL), foscarnet (FOS), Cidofovir, CMX-001, maribavir; acyclovir has no known therapeutic efficacy against CMV and is allowable as standard of care to prevent herpes simplex virus (HSV)
* Prophylactic therapy with CMV immunoglobulin or prophylactic antiviral CMV treatment
* Conditioning regimens 30 days (d) prior to trial participation and up to d28 post-HCT
* Disease-based radiation therapy (not total body irradiation)
* Other investigational product-concurrent enrollment in other clinical trials using any investigational new drug (IND) drugs with unknown effects on CMV or with unknown toxicity profiles is prohibited
* Other medications that might interfere with the evaluation of the investigational product
* Patients with active autoimmune conditions requiting systemic immunosuppressive therapy within the previous 5 years at not eligible
* Patients considered by PIs/protocol team to have a complicated prior therapy or HCT regimen, or who have a low survival probability (e.g., refractory leukemia and/or undergoing 2nd HCT)
* Poor risk disease/disease status including: chronic myeloid leukemia (CML) in blast crisis, acute myeloid leukemia (AML)/acute lymphoblastic leukemia (ALL) beyond 2nd remission, multiple myeloma, and aplastic anemia
* Pregnant women and women who are lactating; breastfeeding should be discontinued if the mother is enrolled on this study
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., social/psychological issues, etc
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Cytomegalovirus (CMV) events | Up to 3 years
  Will include any CMV reactivation (detection of >= 1250 U/mL plasma), low-level reactivation prompting antiviral therapy, or CMV disease (defined by histology) prior to day 100 post-hematopoietic cell transplantation (HCT).

SECONDARY OUTCOMES:
Non-relapse mortality (NRM) | At 100 days post HCT
Severe (grade 3-4) acute graft versus host disease (GVHD) | Up to 3 years
Grade 3-4 adverse events probably/definitely related to the vaccination and modified vaccinia Ankara vector persistence | Up to 3 years
Duration of viremia | Up to 3 years
  The primary statistical analyses will compare vaccine and placebo regarding hazards of CMV events from injection to day 100. Events prior to injection will inform Kaplan Meier estimates for both arms to obtain unbiased estimates of reactivation rates applicable to all transplanted subjects on each arm.
Duration of anti-CMV therapy | Up to 3 years
Peak CMV polymerase chain reaction value | Up to 3 years
Recurrence of CMV viremia | Up to 3 years
Incidence of late CMV reactivation or disease | Up to 3 years
Time to engraftment | Up to 3 years
Incidence of acute GVHD | Up to 3 years
  Will be scored using Keystone consensus criteria. Whenever possible, acute GVHD will be confirmed histologically with microscopic review.
Incidence of chronic GVHD | Up to 3 years
Relapse | Up to 3 years
Non-relapse mortality | Up to 3 years
All-cause mortality | Up to 3 years
Infections | Up to 3 years
Overall survival | Up to 3 years
Levels of CMV-specific T cell immunity | Up to 3 years
  Will also assess immunophenotyping and function.
Natural killer cell function | Up to 3 years
  Will assess cytotoxicity of NK cells against K562 target cell line compared with control (% killing) and cytokine production using flow-cytometry with intra-cellular staining of gamma-interferon and other cytokines (% of NK cells producing these cytokines).

CONTACTS AND LOCATIONS:
Overall Officials: Ryotaro Nakamura, MD, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - Northside Hospital, Atlanta, Georgia
  - Dana-Farber Cancer Institute, Boston, Massachusetts